CLINICAL TRIAL: NCT05303688
Title: Does Preventive Single Dose of Intravenous Dexketoprofen Reduce Pain and Swelling After Orthognathic Surgery? A Prospective, Randomized, Double Blind Clinical Trial
Brief Title: Does Preventive Dexketoprofen Reduce Pain After Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yusuf Nuri Kaba, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Erü Dentistry
Record Dates: First submitted 2022-03-01; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative
Keywords: Preventive analgesia; Pain; Swelling; Orthognathic surgery; Dexketoprofen; 3dMD
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Dexketoprofen Tremetamol (Experimental): 50 mg iv dexketoprofen trometamol (Arveles 50mg/2mL; UFSA, Istanbul, Turkey) were administrated 30 minutes before incision in the treatment group (deksketoprofen trometamol n= 15)
  Interventions: Drug: iv dexketoprofen trometamol (Arveles 50mg/2mL; UFSA, İstanbul, Turkey)
- Drug: Steril Salin (control) (Placebo Comparator): iv sterile saline were administrated 30 minutes before incision in the placebo group (saline n= 15)
  Interventions: Drug: Steril Salin (control)

INTERVENTIONS:
Drug: iv dexketoprofen trometamol (Arveles 50mg/2mL; UFSA, İstanbul, Turkey) — The primary predictor variable was preventive analgesia group. Patients were randomly divided in two groups. 50 mg iv dexketoprofen trometamol (Arveles 50mg/2mL; UFSA, İstanbul, Turkey) were administrated 30 minutes before incision in the treatment group (dexketoprofen trometamol n= 15
  Arms: Drug: Dexketoprofen Tremetamol
Drug: Steril Salin (control) — 30 minutes before incision in the treatment group (dexketoprofen trometamol n= 15) and iv sterile saline were administrated 30 minutes before incision in the placebo group (saline n= 15).
  Arms: Drug: Steril Salin (control)

SUMMARY:
Background The purpose of this study was to evaluate the effect of a single-dose intravenous dexketoprofen administration for preventive analgesia on postoperative pain and reducing swelling in double jaw surgery.

Material and Methods The authors designed a prospective, randomized, and double-blind cohort study. Patients who have Class III malocclusion were randomly divided in two groups. 50 mg intravenous dexketoprofen trometamol were administrated 30 minutes before incision in treatment group, while intravenous sterile saline was administrated 30 minutes before incision in placebo group. The primary predictor variable was treatment group. Primary outcomes were pain, swelling and 24-hour opioid intake. Patient- controlled analgesia with tramadol was given for management of postoperative pain. Other variables were demographic and operation related parameters. Visual analogue scale was used to evaluate postoperative pain. 3dMD Face System (3dMD, USA) was used to measure postoperative swelling. Data were analysed using two independent samples t test and Mann Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study were as follows;
* patients,
* 18-45-year-olds,
* ASA I status,
* Class III malocclusion,
* elective double jaw surgery.

Exclusion Criteria:

* Exclusion criteria were ASA II and above,
* drug allergy,
* liver and kidney failure,
* pregnant or breastfeeding,
* long-term use of pain relievers such as NSAIDs and opioids,
* diabetes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative 1st hours Pain Score on the Visual Analog Scale | postoperative 1st hours
  The postoperative pain was assessed using a 10-cm visual analogue scale (VAS) at postoperative 1st hours. "0" represents least pain, "50" represents moderate pain, and 100 represents maximum pain.
Postoperative 3rd hours Pain Score on the Visual Analog Scale | postoperative 3rd hours.
  The postoperative pain was assessed using a 10-cm visual analogue scale (VAS) at postoperative 3rd hours. "0" represents least pain, "50" represents moderate pain, and 100 represents maximum pain.
Postoperative 6th hours Pain Score on the Visual Analog Scale | postoperative 6th hours.
  The postoperative pain was assessed using a 10-cm visual analogue scale (VAS) at postoperative 6th hours."0" represents least pain, "50" represents moderate pain, and 100 represents maximum pain.
Postoperative 9th hours Pain Score on the Visual Analog Scale | postoperative 9th hours.
  The postoperative pain was assessed using a 10-cm visual analogue scale (VAS) at postoperative 9th hours."0" represents least pain, "50" represents moderate pain, and 100 represents maximum pain.
Postoperative 12th hoursPain Score on the Visual Analog Scale | postoperative 12th hours.
  The postoperative pain was assessed using a 10-cm visual analogue scale (VAS) at postoperative 12th hours. "0" represents least pain, "50" represents moderate pain, and 100 represents maximum pain.
Postoperative 24th hours Pain Score on the Visual Analog Scale | postoperative 24th hours.
  The postoperative pain was assessed using a 10-cm visual analogue scale (VAS) at postoperative 24th hours. "0" represents least pain, "50" represents moderate pain, and 100 represents maximum pain.
3D measure of postoperative swelling | 3D images were taken one (T0) day before surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken 1 (T1) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken3 (T3) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken 7 (T7) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken 14 (T14) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken 21 (T21) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken 30 (T30) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated
3D measure of postoperative swelling | 3D images were taken 90 (T90) day after surgery.
  3dMD Face System (3dMD, ATLANTA, GA, USA) was used for 3D imaging of postoperative swelling. The same clinician took the 3D images from patients in natural head position, maximum intercuspation and eyes open. The 3dMD Vultus Software (3dMD, Atlanta, GA) was used to analyse the images. The 3-month postoperative 3D image (t90) was selected as the reference image to compare with other images. After cutting and customizing the images by anatomical structures, scans t0-t30 were matched to the reference scan t90. The forehead, nasion, tragus, medial and lateral canthus were used for surface matching. After surface matching, the volume difference between the masks was calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Yusuf Nuri Kaba, Kayseri, Melikgazi, Turkey (Türkiye)